CLINICAL TRIAL: NCT02106442
Title: 36-month Special Drug Use Surveillance on Frequency of Bone Fractures With Benet 75 mg Tablets
Brief Title: 36-month Special Drug Use Surveillance on Frequency of Bone Fractures With Sodium Risedronate 75 mg Tablets
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 178-002; JapicCTI-142479 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Osteoporosis
Keywords: Pharmacological therapy
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sodium Risedronate 75 mg: 75 mg of sodium risedronate is administered orally with a sufficient volume (approximately 180 mL) of water once monthly after waking. Participants receive sodium risedronate 75 mg as part of routine medical care.
  Interventions: Drug: Sodium risedronate

INTERVENTIONS:
Drug: Sodium risedronate — Sodium risedronate tablets

SUMMARY:
The purpose of this survey is to evaluate the effectiveness (endpoints: frequency of bone fractures, percent change in bone density, etc.) and safety of administration of sodium risedronate tablets 75 mg for 36 months in osteoporosis patients in daily medical practice.

DETAILED DESCRIPTION:
This special drug use surveillance was designed to evaluate the effectiveness (endpoints: frequency of bone fractures, percent change from baseline in bone density, etc.) and safety of sodium risedronate 75 mg tablets in osteoporosis patients in daily medical practice.

The usual dosage for adult is 75 mg of sodium risedronate administered orally with a sufficient volume (approximately 180 mL) of water once monthly after waking.

ELIGIBILITY:
Inclusion Criteria:

Osteoporosis patients who meet all the following criteria:

1. Patients with 1 to 4 confirmed vertebral body fractures in the T4-L4 region by thoracic and lumbar spine X-ray examination at screening (within 3 months before the start of administration of sodium risedronate 75 mg tablets)
2. Male and postmenopausal female patients aged 50 years or older
3. Ambulatory outpatients

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 148 investigative sites in Japan, from 13 May 2013 to 30 April 2018.
Pre-assignment Details: Participants with a historical diagnosis of osteoporosis were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Sodium Risedronate 75 mg: 75 mg of sodium risedronate was administered orally with a sufficient volume (approximately 180 mL) of water once monthly after waking. Participants received sodium risedronate 75 mg as part of routine medical care.
Period: Overall Study
Arm/Group | Sodium Risedronate 75 mg
Started | 579
Completed | 542
Not Completed | 37
Not completed — Case Report Forms Uncollected | 7
Not completed — Protocol Deviation | 30

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 542
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 541
    (all) | 75.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 479
  Male | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 542
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 304
    (all) | 148.65 (7.88)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 348
    (all) | 50.37 (11.79)
BMI [Mean (Standard Deviation); unit: Kg/meters (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kg/meters (m)^2
    number analyzed (Participants) | 277
    (all) | 22.81 (4.81)
Osteoporosis Class [Count of Participants; unit: Participants]
  Primary Osteoporosis | 481
  Secondary Osteoporosis | 28
  Unknown | 33
Duration of Diagnosis of Osteoporosis [Mean (Standard Deviation); unit: Years] — Mean duration from the first time of diagnosis of osteoporosis to the start of the study was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 462
    (all) | 1.5 (2.8)
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had Predisposition to Hypersensitivity | 32
    Had No Predisposition to Hypersensitivity | 457
    Unknown | 53
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Medical Complications | 453
    Had No Medical Complications | 89
Medical History, Excluding History of Fracture [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had Medical History | 111
    Had No Medical History | 397
    Unknown | 34
Fracture Risk Factor: Medical History of Fracture [Count of Participants; unit: Participants]
  Had Medical History | 305
  Had No Medical History | 212
  Unknown | 25
Fracture Risk Factor: History of Steroid Use, Excluding Steroids for External Use [Count of Participants; unit: Participants]
  Had History of Steroid Use | 35
  Had No History of Steroid Use | 477
  Unknown | 30
Fracture Risk Factor: Parental History of Femur Fracture [Count of Participants; unit: Participants]
  Had Family History of Femur Fracture | 5
  Had No Family History of Femur Fracture | 243
  Unknown | 294
Fracture Risk Factor: Alcohol Classification [Count of Participants; unit: Participants]
  Drank >= 3 Units Daily | 27
  Drank <3 Units Daily | 356
  Unknown | 159
Fracture Risk Factor: Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 324
  Current Smoker | 22
  Ex-Smoker | 21
  Unknown | 175
Previous Medication for Osteoporosis [Count of Participants; unit: Participants]
  Had Previous Medication for Osteoporosis | 201
  Had No Previous Medication for Osteoporosis | 341
Concurrent Medication [Count of Participants; unit: Participants]
  Had Concurrent Medication | 452
  Had No Concurrent Medication | 90
Physical Therapy [Count of Participants; unit: Participants]
  Had Physical Therapy | 178
  Had No Physical Therapy | 364
Other Concurrent Therapy [Count of Participants; unit: Participants] — Other concurrent therapy included diet therapy, exercise therapy, and nerve block.
  Participants
    Had Other Concurrent Therapy | 164
    Had No Other Concurrent Therapy | 378
Back Pain [Count of Participants; unit: Participants]
  Had Back Pain | 346
  Had No Back Pain | 97
  Unknown | 99

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Percentage of Participants With New or Worsening Vertebral Body Fractures
Description: The cumulative data was collected between baseline and Month 36, and reported for the following time points: baseline, Months 6, 12, 18, 24, 30, and 36.
Time Frame: From baseline up to Month 36
Population: Vertebral fractures assessment population; The vertebral fractures assessment population was defined as participants who completed the survey and had evaluable vertebral fractures data at baseline and post-baseline time points. Number analyzed is the number of participants who were evaluable at each time point.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 328
Percentage of Participants
  Month 6: number analyzed (Participants) | 254
  Month 6 | 5.43 [3.36 to 8.72]
  Month 12: number analyzed (Participants) | 227
  Month 12 | 7.35 [4.85 to 11.06]
  Month 18: number analyzed (Participants) | 192
  Month 18 | 7.80 [5.20 to 11.64]
  Month 24: number analyzed (Participants) | 172
  Month 24 | 8.82 [5.97 to 12.93]
  Month 30: number analyzed (Participants) | 142
  Month 30 | 9.97 [6.84 to 14.43]
  Month 36: number analyzed (Participants) | 69
  Month 36 | 12.58 [8.61 to 18.18]

2. Secondary Outcome: Cumulative Percentage of Participants With Non-Vertebral Body Fractures
Description: as for outcome 1
Time Frame: From baseline up to Month 36
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available. Number analyzed is the number of participants who were evaluable at each time point.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 535
Percentage of Participants
  Month 6: number analyzed (Participants) | 401
  Month 6 | 1.72 [0.86 to 3.41]
  Month 12: number analyzed (Participants) | 348
  Month 12 | 2.78 [1.58 to 4.86]
  Month 18: number analyzed (Participants) | 284
  Month 18 | 3.40 [2.01 to 5.71]
  Month 24: number analyzed (Participants) | 259
  Month 24 | 4.11 [2.51 to 6.69]
  Month 30: number analyzed (Participants) | 218
  Month 30 | 6.15 [3.99 to 9.43]
  Month 36: number analyzed (Participants) | 133
  Month 36 | 6.59 [4.31 to 10.01]

3. Secondary Outcome: Cumulative Percentage of Participants With Femur Fractures
Description: as for outcome 1
Time Frame: From baseline up to Month 36
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 535
Percentage of Participants
  Month 6: number analyzed (Participants) | 407
  Month 6 | 0.19 [0.03 to 1.35]
  Month 12: number analyzed (Participants) | 355
  Month 12 | 0.46 [0.11 to 1.84]
  Month 18: number analyzed (Participants) | 290
  Month 18 | 0.78 [0.25 to 2.46]
  Month 24: number analyzed (Participants) | 266
  Month 24 | 1.14 [0.42 to 3.08]
  Month 30: number analyzed (Participants) | 228
  Month 30 | 1.14 [0.42 to 3.08]
  Month 36: number analyzed (Participants) | 139
  Month 36 | 1.58 [0.64 to 3.88]

4. Secondary Outcome: Percent Change From Baseline in Mean Lumbar Spine (L2-L4) Bone Mineral Density (BMD) at Final Assessment (up to Month 36)
Description: BMD was measured by dual-energy X-ray absorptiometry.
Time Frame: Baseline and final assessment (up to Month 36)
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available. Number analyzed is the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 122
Percent Change | 6.848 (8.971)

5. Secondary Outcome: Percent Change From Baseline in Femur Neck BMD at Final Assessment (up to Month 36)
Description: BMD was measured by dual-energy X-ray absorptiometry.
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 93
Percent Change | 1.067 (6.757)

6. Secondary Outcome: Percent Change From Baseline in Total Proximal Femur BMD at Final Assessment (up to Month 36)
Description: BMD was measured by dual-energy X-ray absorptiometry.
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 103
Percent Change | 1.496 (6.841)

7. Secondary Outcome: Percent Change From Baseline in Radius BMD at Final Assessment (up to Month 36)
Description: BMD was measured by dual-energy X-ray absorptiometry.
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 119
Percent Change | 3.498 (10.608)

8. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Type 1 Collagen Cross-linked N-telopeptide (NTX) at Final Assessment (up to Month 36)
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 21
Percent Change | -15.756 (26.386)

9. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Tartrate-resistant Acid Phosphatase 5b (TRACP-5b) at Final Assessment (up to Month 36)
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 97
Percent Change | -15.539 (130.961)

10. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Bone-type Alkaline Phosphatase (BAP) at Final Assessment (up to Month 36)
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 22
Percent Change | -20.023 (23.160)

11. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Procollagen 1 N-terminal Peptide (P1NP) at Final Assessment (up to Month 36)
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 51
Percent Change | -40.838 (40.776)

12. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Urinary Type 1 Collagen Cross-linked N-telopeptide (NTX) at Final Assessment (up to Month 36)
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 33
Percent Change | -25.285 (62.112)

13. Secondary Outcome: Change From Baseline in Height at Final Assessment (up to Month 36)
Time Frame: Baseline and final assessment (up to Month 36)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 164
Centimeter | -0.82 (1.35)

14. Secondary Outcome: Number of Participants Who Had Lumbar Backache at Final Assessment (up to Month 36)
Time Frame: Final assessment (up to Month 36)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 376
Participants | 116

15. Secondary Outcome: Number of Participants Who Had One or More Adverse Drug Reactions
Description: Adverse drug reaction refers to adverse events related to the administered drug.
Time Frame: Up to Month 36
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 542
Participants | 57

ADVERSE EVENTS:
Time Frame: Up to Month 36
Description: At each visit the investigator had to document any occurrence of adverse events (AEs) and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment. Only adverse drug reactions (ADRs) were collected and reported on safety results sections here.
Arm/Group | Sodium Risedronate 75 mg
All-Cause Mortality (participants affected / at risk) | 0/542
Serious Adverse Events (participants affected / at risk) | 4/542
Other Adverse Events (participants affected / at risk) | 7/542
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Risedronate 75 mg (N=542)
Toothache (Gastrointestinal disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hospitalisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Risedronate 75 mg (N=542)
Nausea (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT02106442/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT02106442/SAP_001.pdf